CLINICAL TRIAL: NCT06389136
Title: A Phase 3b/4 Randomized, Open-label, Efficacy Assessor-Blinded Study, to Evaluate the Efficacy and Safety of Upadacitinib for the Treatment of Adult Subjects With Moderate to Severe Atopic Dermatitis and Inadequate Response to Dupilumab (SWITCH-UP)
Brief Title: A Study of Upadacitinib in Adult Participants With Moderate-to-Severe Atopic Dermatitis and Inadequate Response to Dupilumab
Acronym: Switch-Up
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M24-601; 2025-523347-35 (Other: EU CT)
Record Dates: First submitted 2024-04-25; First posted 2024-04-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: Upadacitinib; Rinvoq; ABT-494
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib; dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Period 1: Upadacitinib Open Label Treatment (Experimental): Participants randomly assigned to receive Upadacitinib 15mg tablet once per day.
  Based on clinical response, participants randomized to Upadacitinib 15mg may have their dose increased to Upadacitinib 30mg starting at Week 2.
  Interventions: Drug: Upadacitinib 15mg Dose; Drug: Upadacitinib 30mg Dose
- Period 1: Dupilumab Open Label Treatment (Experimental): Participants randomly assigned to receive Dupilumab 300mg SC injection once every other week for 8 weeks.
  Interventions: Drug: Dupilumab 300mg Dose
- Period 2 Open Label: Upadacitinib < EASI 75 response (Experimental): Participants that were receiving Upadacitinib 15mg or 30mg and completed Period 1, will be allocated or continue to receive oral doses of Upadacitinib 30mg in Period 2 with a clinical response of < EASI 75 at Week 8
  Interventions: Drug: Upadacitinib 30mg Dose
- Period 2 Open Label: Upadacitinib ≥ EASI 75 Response (Experimental): Participants that were receiving Upadacitinib 15mg or 30mg and completed Period 1, will continue to receive the same oral doses of Upadacitinib in Period 2 with a clinical response of ≥ EASI 75 at Week 8
  Interventions: Drug: Upadacitinib 15mg Dose; Drug: Upadacitinib 30mg Dose
- Period 2 Open Label: Dupilumab ≥ EASI 75 Response (Experimental): Participants that were receiving Dupilumab 300mg and completed Period 1, will continue to receive Dupilumab 300mg SC injection in Period 2 with a clinical response of ≥ EASI 75 at Week 8
  Interventions: Drug: Dupilumab 300mg Dose
- Period 2 Open Label Period: Dupilumab < EASI 75 Response (Experimental): Participants that were receiving Dupilumab 300mg SC injections and completed Period 1, will receive oral doses of Upadacitinib 15mg in Period 2 with a clinical response of < EASI 75 at Week 8
  Interventions: Drug: Upadacitinib 15mg Dose

INTERVENTIONS:
Drug: Upadacitinib 15mg Dose — Oral tablet
  Other Names: ABT-494; RINVOQ
  Arms: Period 1: Upadacitinib Open Label Treatment; Period 2 Open Label Period: Dupilumab < EASI 75 Response; Period 2 Open Label: Upadacitinib ≥ EASI 75 Response
Drug: Dupilumab 300mg Dose — Subcutaneous (SC) injection
  Arms: Period 1: Dupilumab Open Label Treatment; Period 2 Open Label: Dupilumab ≥ EASI 75 Response
Drug: Upadacitinib 30mg Dose — Oral tablet
  Other Names: ABT-494; RINVOQ
  Arms: Period 1: Upadacitinib Open Label Treatment; Period 2 Open Label: Upadacitinib < EASI 75 response; Period 2 Open Label: Upadacitinib ≥ EASI 75 Response

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. Therapies spread over the skin may not be enough to control the AD in trial participants who require systemic anti-inflammatory treatment. This study aims to provide data on the efficacy and safety of upadacitinib at different doses in adult participants with moderate to severe AD.

Upadacitinib is an approved drug for the treatment of moderate to severe atopic dermatitis (AD). This study is conducted in 2 periods. During Period 1, participants are randomly assigned into 1 of 2 groups called treatment arms to receive upadacitinib 15mg or dupilumab 300mg. Based on the participants response to upadacitinib 15mg, they may have their dose increased to upadacitinib 30mg after 2 weeks. In Period 2, participants that completed Period 1 will either remain on their assigned dose or be reassigned to a different dose based on their Eczema Area and Severity Index (EASI) response. Approximately 200 adult participants ages 18 to less than 64 with moderate to severe AD who are current users of dupilumab and had a history of inadequate response to dupilumab will be enrolled at up to 130 sites worldwide.

The study is comprised of a 35-day Screening Period, an 8-week Open-Label Period 1 and a 24-week Open-Label Period 2 for participants that completed Period 1. Participants will receive upadacitinib oral tablets once daily or dupilumab subcutaneous (SC) injection every other week for 32 weeks and followed for 30 days.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Chronic AD with onset of symptoms at least 3 years prior to Baseline and subject meets Hanifin and Rajka criteria.
* Participant meets all the following disease activity criteria at Baseline Visit:

  * Eczema Area and Severity Index (EASI) score >= 12;
  * validated Investigator´s Global Assessment for AD (vIGA-AD) score >= 3;
  * Body surface area (BSA) involvement of >= 10% in a majority of subjects (>= 50% of the overall study population)
  * Baseline weekly average of daily Worst Pruritus-Numerical Rating Scale (WP-NRS) >= 4. Note: The Baseline weekly average of daily WP-NRS will be calculated from the 7 consecutive days immediately preceding the Baseline Visit. A minimum of 4 daily scores out of the 7 days is needed.
  * Inadequate response to dupilumab treatment after at least 4 months of current use.
  * Particpant has applied a topical emollient (an additive-free, bland emollient moisturizer) twice daily for at least 7 days before the Baseline Visit and for the duration of the study. Note: Subject may use prescription moisturizers or moisturizers containing ceramide, urea, filaggrin degradation products or hyaluronic acid if such moisturizers were initiated before the Screening visit.

Exclusion Criteria:

* Meeting any of the following conditions at Baseline:

  * Other active skin diseases or skin infections (bacterial, fungal, or viral) requiring systemic treatment within 4 weeks of the Baseline Visit or would interfere with assessment of AD lesions;
  * Two or more past episodes of herpes zoster, or one or more episodes of disseminated herpes zoster;
  * One or more past episodes of disseminated herpes simplex (including eczema herpeticum);
  * HIV infection defined as confirmed positive anti- HIV Ab test;
  * Participants with current or past history of infection including, Evidence of Hepatitis B virus (HBV) or Hepatitis C virus (HCV);
  * Active TB or meet TB exclusionary parameters (specific requirements for TB testing are provided in the operations manual);
  * For Japan: Positive result of beta-D-glucan (screening for Pneumocystis jirovecii infection) or two consecutive indeterminate results of beta-D-glucan during the Screening Period;
  * Active infection(s) requiring treatment with intravenous anti-infectives within 30 days, or oral/intramuscular anti-infectives within 14 days prior to the Baseline Visit;
  * Chronic recurring infection and/or active viral infection that, based on the investigator's clinical assessment, makes the subject an unsuitable candidate for the study;
  * COVID-19 infection: In subjects who tested positive for COVID-19, at least 5 days must have passed between a COVID-19 positive test result and the Baseline visit of asymptomatic subjects. Subjects with mild/moderate COVID-19 infection can be enrolled if fever is resolved without use of antipyretics for 24 hours and other symptoms improved, or if 5 days have passed since the COVID-19 positive test result (whichever comes last). Subjects may be rescreened if deemed appropriate by the investigator based upon the subject's health status.
* At Baseline any of the following medical diseases or disorders:

  * Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting, and aorto-coronary bypass surgery or venous thromboembolism;
  * Any unstable clinical condition which, in the opinion of the investigator would put the subject at risk by participating in the protocol;
  * Diagnosed active parasitic infection, suspected or high risk of parasitic infection unless clinical (and if necessary) laboratory assessment have ruled out active infection before randomization;
  * History of an organ transplant which requires continued immunosuppression;
  * History of an allergic reaction or significant sensitivity to constituents of the study drug (and its excipients) and/or other products in the same class;
  * History of GI perforation (other than due to appendicitis or mechanical injury), diverticulitis, or significantly increased risk for GI perforation per investigator judgment;
  * Conditions that could interfere with drug absorption including but not limited to short bowel syndrome or gastric bypass surgery including sleeve gastrectomy; subjects with a history of gastric banding/segmentation are not excluded;
  * History of malignancy except for successfully treated NMSC or localized carcinoma in situ of the cervix.

Ages: 18 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Participants who achieve at least a 90% reduction in Eczema Area and Severity Index from Baseline (EASI 90) | At Week 8
  The EASI is a validated measure used to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points.

SECONDARY OUTCOMES:
Percentage of participants who achieve a Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) | At Week 8
  Worst Pruritus NRS (WP-NRS) is a validated single self-reported measure where patients rate the worst level of itching they have experienced over the past 24 hours on a scale from 0 (no itching) to 10 (worst itching imaginable)
Participants who simultaneous achieve at least a 90% reduction in Eczema Area and Severity Index from Baseline (EASI 90) and Worst Pruritus Numerical Rating Scale of 0 or 1 (WP-NRS 0/1) | At Week 8
  The EASI is a validated measure used to assess the severity and extent of AD. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) are each assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe). In addition, the area of AD involvement is assessed as a percentage by body area of head, trunk (including the genital area), upper extremities, and lower extremities (including the buttocks), and converted to a score of 0 to 6. In each body region, the area is expressed as 0, 1 (1% to 9%), 2 (10% to 29%), 3 (30% to 49%), 4 (50% to 69%), 5 (70% to 89%), or 6 (90% to 100%). The EASI score ranges from 0-72 points with an MCID of 6.6 points. Worst Pruritus NRS (WP-NRS) is a validated single self-reported measure where patients rate the worst level of itching they have experienced over the past 24 hours on a scale from 0 (no itching) to 10 (worst itching imaginable)
Percentage of participants achieving worst pruritus numerical rating scale (WP-NRS) 0/1 | At Week 4
  Worst Pruritus NRS (WP-NRS) is a validated single self-reported measure where patients rate the worst level of itching they have experienced over the past 24 hours on a scale from 0 (no itching) to 10 (worst itching imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (104):
- United States (74):
  - Clinical Trials Institute - Northwest Arkansas /ID# 267290, Fayetteville, Arkansas
  - Private Practice - Dr. Tooraj Raoof /ID# 263849, Encino, California
  - First OC Dermatology /ID# 263349, Fountain Valley, California
  - NorCal Medical Research /ID# 278397, Greenbrae, California
  - Allergy & Asthma Associates of Southern California - Mission Viejo /ID# 266574, Mission Viejo, California
  - Dermatologist Medical Group of North County- Profound Research /ID# 266512, Oceanside, California
  - Stanford University School of Medicine - Redwood City /ID# 263776, Redwood City, California
  - Integrative Skin Science and Research /ID# 264537, Sacramento, California
  - West Dermatology La Jolla /ID# 265014, San Diego, California
  - Clinical Trials Research Institute /ID# 263846, Thousand Oaks, California
  - Yale University School of Medicine /ID# 263836, New Haven, Connecticut
  - Clearlyderm Dermatology - West Boca /ID# 264923, Boca Raton, Florida
  - Skin Care Research Boca Raton /ID# 263733, Boca Raton, Florida
  - Apex Clinical Trials /ID# 263747, Brandon, Florida
  - TrueBlue Clinical Research /ID# 265037, Brandon, Florida
  - Life Clinical Trials /ID# 267195, Coral Springs, Florida
  - Revival Research - Doral /ID# 263541, Doral, Florida
  - Skin Care Research - Hollywood /ID# 263739, Hollywood, Florida
  - Solutions Through Advanced Research /ID# 263392, Jacksonville, Florida
  - GSI Clinical Research, LLC /ID# 263760, Margate, Florida
  - Research Associates of South Florida /ID# 267291, Miami, Florida
  - International Dermatology Research /ID# 264961, Miami, Florida
  - Sullivan Dermatology /ID# 263537, Miami, Florida
  - Lenus Research and Medical Group /ID# 263779, Miami, Florida
  - Quality Research of South Florida /ID# 266496, Miami Lakes, Florida
  - Global Clinical Professionals (GCP) /ID# 266474, St. Petersburg, Florida
  - Skin Care Research - Tampa /ID# 263750, Tampa, Florida
  - Alliance Clinical Research of Tampa /ID# 264531, Tampa, Florida
  - Encore Medical Research - Weston /ID# 278491, Weston, Florida
  - Centricity Research Columbus Dermatology /ID# 266529, Columbus, Georgia
  - Cleaver Medical Group Dermatology /ID# 263788, Dawsonville, Georgia
  - Georgia Skin & Cancer Clinic /ID# 267199, Savannah, Georgia
  - Treasure Valley Medical Research /ID# 263738, Boise, Idaho
  - DeNova Research /ID# 264513, Chicago, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 264983, Chicago, Illinois
  - Dawes Fretzin, LLC /ID# 264534, Indianapolis, Indiana
  - Options Research Group /ID# 264564, West Lafayette, Indiana
  - Dermatology Specialists Research (DS Research) - Kentucky /ID# 263388, Louisville, Kentucky
  - Velocity Clinical Research at The Dermatology Clinic - Baton Rouge /ID# 267169, Baton Rouge, Louisiana
  - Boston Specialists /ID# 265810, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 263703, Boston, Massachusetts
  - Beacon Clinical Research /ID# 263843, Quincy, Massachusetts
  - Great Lakes Research Group - Bay City /ID# 263535, Bay City, Michigan
  - Henry Ford Medical Center - New Center One /ID# 263522, Detroit, Michigan
  - Onyx Clinical Research - Flint - South Linden Road /ID# 267773, Flint, Michigan
  - MediSearch Clinical Trials /ID# 263579, Saint Joseph, Missouri
  - Physician Research Collaboration, LLC /ID# 263583, Lincoln, Nebraska
  - Skin Specialists /ID# 263345, Omaha, Nebraska
  - Skin Cancer and Dermatology Institute - Reno /ID# 263771, Reno, Nevada
  - Dartmouth Hitchcock Medical Center - Old Etna Road /ID# 263840, Lebanon, New Hampshire
  - Forest Hills Dermatology Group @ Union Turnpike /ID# 263755, Kew Gardens, New York
  - Equity Medical, LLC /ID# 265814, New York, New York
  - Weill Cornell Medicine /ID# 265793, New York, New York
  - Piedmont Plastic Surgery and Dermatology /ID# 266545, Huntersville, North Carolina
  - Vital Prospects Clinical Research Institute - Tulsa /ID# 263645, Tulsa, Oklahoma
  - Oregon Health and Science University /ID# 263736, Portland, Oregon
  - Dermatology Partners /ID# 264972, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center /ID# 264526, Pittsburgh, Pennsylvania
  - Dermatology Associates of Plymouth Meeting /ID# 267286, Plymouth Meeting, Pennsylvania
  - Medical University of South Carolina /ID# 263655, Charleston, South Carolina
  - ADCS - Spartanburg /ID# 267185, Spartanburg, South Carolina
  - Health Concepts /ID# 263383, Rapid City, South Dakota
  - Arlington Research Center, Inc /ID# 263665, Arlington, Texas
  - Orion Clinical Research /ID# 263658, Austin, Texas
  - Bellaire Dermatology Associates /ID# 263794, Bellaire, Texas
  - Studies in Dermatology LLC /ID# 263335, Cypress, Texas
  - Dermatology Treatment and Research Center /ID# 265812, Dallas, Texas
  - Modern Research Associates /ID# 263852, Dallas, Texas
  - The Dermatology Institute of South Texas /ID# 267332, McAllen, Texas
  - Texas Dermatology Research Center /ID# 264528, Plano, Texas
  - Stride Clinical Research /ID# 267331, Sugar Land, Texas
  - The Woodlands Dermatology Associates /ID# 266547, The Woodlands, Texas
  - Dermatology Associates of Tyler /ID# 264980, Tyler, Texas
  - West Virginia Research Institute - Morgantown /ID# 264930, Morgantown, West Virginia
- Canada (5):
  - Dermatology Research Institute - Blackfoot Trail /ID# 270450, Calgary, Alberta
  - Stratica Medical /ID# 270466, Edmonton, Alberta
  - York Dermatology Clinic & Research Centre /ID# 278847, Richmond Hill, Ontario
  - Centre de Recherche dermatologique du Quebec Metropolitain /ID# 277564, Québec, Quebec
  - Centre de Recherche Saint-Louis /ID# 271083, Québec, Quebec
- Colombia (4):
  - Centro de Inmunología y Genética CIGE SAS /ID# 266200, Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe SAS - Circaribe SAS /ID# 265088, Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y especialidades Medicas S.A.S- CIREEM /ID# 265092, Bogotá, Cundinamarca
  - Unidad Integral de Endocrinologia (UNIENDO) /ID# 266970, Bogotá, Cundinamarca
- Japan (10):
  - Ichinomiya Municipal Hospital /ID# 265068, Ichinomiya, Aichi-ken
  - Takeoka Dermatology Clinic /ID# 264055, Marugame, Kagawa-ken
  - Kawasaki Medical School Hospital /ID# 266164, Kurashiki, Okayama-ken
  - Dokkyo Medical University Hospital /ID# 265431, Mibu, Tochigi
  - Ogikubo Hospital /ID# 278350, Suginami-Ku, Tokyo
  - Tachikawa Dermatology Clinic /ID# 271912, Tachikawa-shi, Tokyo
  - Yamanashi Prefectural Central Hospital /ID# 278052, Kofu, Yamanashi
  - Katahira Dermatology Urology Clinic /ID# 264403, Kagoshima
  - NTT Medical Center Tokyo /ID# 265104, Tokyo
  - Teikyo University Hospital /ID# 265126, Tokyo
- Puerto Rico (6):
  - SCB Research Center /ID# 263217, Bayamón
  - Private Practice - Dr. Samuel Sanchez /ID# 263199, Caguas
  - Private Practice - Dr. Alma Cruz /ID# 263216, Carolina
  - Clinical Research Puerto Rico /ID# 263197, San Juan
  - GCM Medical Group, PSC /ID# 263218, San Juan
  - CMRC Headlands LLC /ID# 267163, San Juan
- South Korea (5):
  - Korea University Ansan Hospital /ID# 263330, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 263331, Bucheon-si, Gyeonggido
  - Ajou University Hospital /ID# 263328, Suwon, Gyeonggido
  - Seoul National University Hospital /ID# 263329, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 263327, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-601